CLINICAL TRIAL: NCT02537145
Title: Do-It-Yourself Health Monitoring and Simulation of Health in Pregnant Women - Pilot Study
Brief Title: PregnanT Moms Measure - Do-It-Yourself Health Monitoring and Simulation of Health in Pregnant Women
Acronym: oPTiMuM
Status: Terminated | Type: Observational
Why Stopped: Not enough obese subjects could be recruited.
Sponsor: W.J. Pasman (Other)
Collaborators: Spaarne Gasthuis (Other)
Responsible Party: Sponsor-Investigator, W.J. Pasman, Consultant Clinical Trials, TNO
Organization: TNO (Other)
Other Study IDs: P9624
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Pregnancy; Obesity
Keywords: compliance; do-it-yourself methodology; pilot; human microbiome
MeSH Terms: conditions — Obesity; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Finger-prick-blood for dried blood spots will be performed for oral glucose tolerance tests (insuline/c-peptide response profile) and determining protein and lipid metabolism as well as HbA1c.
  Finger-prick-blood for measurement of glucose and cholesterol using do-it-yourself devices.
  Saliva and fecal samples for determining gut and oral microbiota (bacteria) by DNA sequencing of bacterial marker genes present in fecal and saliva samples.
  Hair sample for determining cortisol concentrations over time.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese pregnant women: 20 obese pregnant women (BMI ≥ 30)
- Lean pregnant women: 20 lean pregnant women (BMI 18,5 - 25)

SUMMARY:
The aim of this pilot study is to determine the feasibility of Do-It-Yourself studies in pregnant women to detect changes in health parameters by assessing compliance and user experiences of participants. Besides, the measured health will be analysed to increase insight in physiological development in pregnant women.

DETAILED DESCRIPTION:
The study is designed as an open, parallel, do-it-yourself, explorative, two-group study. Subjects are women who are pregnant for approximately 3 months at the start of the study. Subjects will be included between week 12 and 15 of their pregnancy (T=-1). Week 16 is the start of the study (T=0). In the first group obese pregnant women (BMI ≥ 30) will be included; the second group will consist of lean pregnant women (BMI 18,5 - 25).

The women will be requested to assess physiological parameters at regular intervals from three months pregnancy until giving birth (week 40). The assessment after giving birth, until three months after giving birth (total study duration of approximately nine months), is optional.

Health parameters are known to be subject to change in pregnant women; the self-monitoring devices should be able to show these changes. Included subjects will be provided with the do-it-yourself devices, manuals and the study protocol. During the nine-month study, the subjects will use these do-it-yourself devices to self-monitor multiple health parameters in an at-home setting. They will be reminded to perform these tests via SMS. There are two frequency intervals defined (two week interval and eight week interval).

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant between 12-15 weeks at the start of the study;
2. Healthy as assessed by the Health and Lifestyle questionnaire (P9624 F02);
3. Body mass index:

   * BMI 18,5 - 25 for the lean group
   * BMI ≥ 30 for the obese group;
4. Able to use self-monitoring devices;
5. Voluntary participation;
6. Having given written informed consent;
7. Willing to comply with study procedures;
8. Willingness to share pseudonymised data on measured health parameters with external parties that provide the measuring devices (including MijnEetmeter, Moves and NRC) for reasons of synchronisation with the study database;
9. Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data by TNO;
10. Have internet access at home;
11. Subjects should own a Smartphone with Bluetooth that runs either a recent version of iOS or Android.

Exclusion Criteria:

1. Use of concomitant medication;
2. Having a history of medical or surgical events that may significantly affect the study outcome, including physical limitations or cardio-vascular events;
3. Having a (history of a) medical condition that might significantly affect the study outcome as judged by the principal investigator and health and life style questionnaire. This includes diabetes type 1 or 2, gastrointestinal dysfunction, diseases related to inflammation, or a psychiatric disorder;
4. Hypertension: systolic blood pressure >160 mmHg, diastolic blood pressure >90 mmHg;
5. Having a pacemaker;
6. Previous pregnancy with medical issues (e.g. pre-eclampsia);
7. Reported slimming or medically prescribed diet;
8. Physical, mental or practical limitations in using computerized systems;
9. Alcohol consumption > 14 units (drinks)/week;
10. Smoking;
11. Reported unexplained weight loss or gain of > 2 kg in the three months prior to the pre-study screening / pregnancy;
12. Recent blood donation (<1 month prior to the start of the study);
13. Not willing to give up blood donation during the study;
14. Personnel of TNO and their partner.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of 40 women who are between 12 and 15 weeks pregnant at the time of inclusion in the study. In this study, two groups will be compared: 20 obese pregnant women (BMI ≥ 30) and 20 lean pregnant women (BMI 18,5 - 25).
  All pregnant women will be from Dutch descent (Dutch nationality and culture).
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
compliance (percentage of complete datasets) | end of study (3 months after giving birth)
  as a measure of the potential of DIY-monitoring in pregnant women
Capability of and burden for participants of the use of DIY tools | end of study (3 months after giving birth)
  as assessed by a questionnaire on user-experience with do-it-yourself devices in an at-home setting

SECONDARY OUTCOMES:
fasting blood glucose | at enrollment (between w12-15 of pregnancy), baseline (w16 of pregnancy), w18, 20, 22, 24, 26, 28, 30, 32, 34, 36, 38, 40 of pregnancy; optionally after delivery in w42, 44, 46, 48, 50, 52
  as measured using a do-it-yourself glucose meter after an overnight fast
body weight | at enrollment (between w12-15 of pregnancy), baseline (w16 of pregnancy), w18, 20, 22, 24, 26, 28, 30, 32, 34, 36, 38, 40 of pregnancy; optionally after delivery in w42, 44, 46, 48, 50, 52
  as measured by a smart-scale
physical activity (calories burned, minutes of physical activity, number of steps) | at enrollment (between w12-15 of pregnancy), baseline (w16 of pregnancy), w18, 20, 22, 24, 26, 28, 30, 32, 34, 36, 38, 40 of pregnancy; optionally after delivery in w42, 44, 46, 48, 50, 52
  participants continuously wear the activity tracker during the day for the whole week in each of the above mentioned measurement-weeks
blood pressure (diastolic, systolic, heart rate) | at enrollment (between w12-15 of pregnancy), baseline (w16 of pregnancy), w18, 20, 22, 24, 26, 28, 30, 32, 34, 36, 38, 40 of pregnancy; optionally after delivery in w42, 44, 46, 48, 50, 52
  as measured with a do-it-yourself blood pressure meter
GPS location | measured continuously during the entire study
  measured with an app that will be installed on the Smartphone of the participant at enrollment in the study
Cholesterol (total cholesterol, HDL, LDL, triglycerides, cholesterol/HDL-ratio) | at enrollment (between w12-15 of pregnancy), baseline (w16 of pregnancy), w24, 32, 40 of pregnancy; optionally after delivery in w52
  measured using a do-it-yourself cholesterol meter
oral glucose tolerance test (glucose, insulin, c-peptide) | baseline (w16 of pregnancy), w24, 32, 40 of pregnancy; optionally after delivery in w52
  in week 16 the test will be done in a clinical setting; the other tests will be done at home by the participants
fecal and salivary microbiota composition | at enrollment (between w12-15 of pregnancy), baseline (w16 of pregnancy), w24, 32, 40 of pregnancy; optionally also in w18, 27 and 36, and after delivery in w44, 48 and 52
  using do-it-yourself sample collection kits (at home by participants; samples will be send to the lab)
dried blood spots for HbA1c, fatty acids and blood biomarkers | at enrollment (between w12-15 of pregnancy), baseline (w16 of pregnancy), w24, 32, 40 of pregnancy; optionally after delivery in w52
  do-it-yourself using finger-prick and blood spot collection cards that can be send to the lab.
cortisol in hair | at the end of the study (3 months after delivery; week 52)
  measured by taking a hair sample that is send to the lab
food intake as measured by a web-application | at enrollment (between w12-15 of pregnancy), baseline (w16 of pregnancy), w24, 32, 40 of pregnancy; optionally after delivery in w52
  in each measurement week, participants will register their food intake on two week days and one weekend day
cognition | at enrollment (between w12-15 of pregnancy), baseline (w16 of pregnancy), w24, 32, 40 of pregnancy; optionally after delivery in w52
  using online cognition tests (on a study portal)
Groninger Sleep Scale | at enrollment (between w12-15 of pregnancy), baseline (w16 of pregnancy), w24, 32, 40 of pregnancy; optionally after delivery in w52
  online; can be accessed via the study portal
Vita16 - vitality questionnaire | at enrollment (between w12-15 of pregnancy), baseline (w16 of pregnancy), w24, 32, 40 of pregnancy; optionally after delivery in w52
  online; can be accessed via the study portal
visual analogue scales for general health | at enrollment (between w12-15 of pregnancy), baseline (w16 of pregnancy), w24, 32, 40 of pregnancy; optionally after delivery in w52
  online; can be accessed via the study portal

CONTACTS AND LOCATIONS:
Overall Officials: Marlies A van Houten, Dr., Principal Investigator — Spaarne Gasthuis
Locations (1):
- Spaarne Gasthuis, Hoofddorp, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided